CLINICAL TRIAL: NCT07092085
Title: An Artificial Intelligence-Based Screening Tool to Detect Psychological Distress
Brief Title: AI-Powered Mental Health Screening in University Students
Status: Completed | Type: Observational
Sponsor: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Kang Zhang, Professor, The Eye Hospital of Wenzhou Medical University
Other Study IDs: Mental Health
Record Dates: First submitted 2025-07-10; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Mental Disease
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Control: without mental healthy problem
  Interventions: Diagnostic Test: AI model
- Mental Diseases: with mental problem, such as depression, OCD
  Interventions: Diagnostic Test: AI model

INTERVENTIONS:
Diagnostic Test: AI model — An AI model provides an objective and rapid assessment of potential mental health risks in students by holistically analyzing their facial expressions, vocal characteristics, and linguistic content from data.

SUMMARY:
The goal of this observational study is to test an artificial intelligence (AI) tool that can help screen for mental health risks . The main questions it aims to answer are:

Can an AI model that analyzes a person's voice, facial expressions, and language accurately identify students who may be at high risk for mental health conditions, such as depression or OCD?

How accurate is the AI model when compared to results from standard mental health questionnaires?

Participants will be asked to:

Complete a standard mental health questionnaire.

Provide consent for their data to be used in the research.

Participate in a recorded session to collect video and audio data for the AI model to analyze.

DETAILED DESCRIPTION:
This large-scale, multi-center observational study aims to develop and validate a novel artificial intelligence (AI) model for the early and objective screening of mental health risks, such as depression and OCD, in university students. The model will be trained and internally validated on multimodal data (including vocal, facial, and linguistic features) from a large student cohort. A subsequent neuroscience sub-study will explore the neurobiological correlates of the AI-identified risk levels using electroencephalography (EEG) and functional magnetic resonance imaging (fMRI) to establish biological validity. The primary outcome is to assess the final model's diagnostic accuracy, quantified by its sensitivity, specificity, and AUC, with the ultimate goal of providing a scalable and efficient early warning tool to facilitate timely clinical intervention for university populations.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled as a student at a participating university.
* Age between 14 and 40 years, inclusive.
* Willing and able to provide written informed consent.
* Fluent in the language required for the study.

Exclusion Criteria:

* Inability to provide video or audio data of sufficient quality for analysis.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population comprises a large cohort of students recruited from multiple universities. Participants will be included in the main phase for AI model development. Additionally, a sub-group of students will be selected based on their mental health risk levels (e.g., for depression or OCD) to participate in a subsequent neuroscience sub-study.
Sampling Method: Non-Probability Sample
Enrollment: 17386 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
AUROC | through study completion, an average of 1 year
  Area Under the Receiver Operating Characteristic Curve
Specificity of the AI Model for Mental Health Screening | through study completion, an average of 1 year
  The ability of the AI model to correctly identify students without significant psychological distress. It will be calculated as the percentage of participants correctly classified as 'low-risk' by the AI model compared to a 'gold standard' classification

SECONDARY OUTCOMES:
Positive and Negative Predictive Values | through study completion, an average of 1 year
Correlation Between AI-Identified Risk Scores and Neurobiological Markers | through study completion, an average of 1 year
  To assess the biological validity of the AI model, the model's output will be correlated with specific neurobiological markers obtained from a sub-study. The correlation will be assessed using a Pearson correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No